CLINICAL TRIAL: NCT07037901
Title: A Phase 2b, Multicenter, Randomized, Double-blinded, Placebo-controlled, Parallel-group, Dose-finding Study to Evaluate the Efficacy and Safety of IMG-007 in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Efficacy and Safety of IMG-007 in Adult Participants With Moderate-to-Severe Atopic Dermatitis
Acronym: ADAPTIVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inmagene LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IMG-007-203
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Atopic Dermatitis; Atopic Dermatitis Eczema; Eczema
Keywords: IMG-007; Atopic Dermatitis; Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases; Dermatologic Agents
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases; Immune System Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IMG-007 dose 1 (Experimental): Subcutaneous injection as per protocol.
  Interventions: Drug: IMG-007
- IMG-007 dose 2 (Experimental): Subcutaneous injection as per protocol.
  Interventions: Drug: IMG-007
- IMG-007 dose 3 (Experimental): Subcutaneous injection as per protocol.
  Interventions: Drug: IMG-007
- Placebo Crossover (Placebo Comparator): Subcutaneous placebo injection as per protocol. At crossover, IMG-007 subcutaneous injection as per protocol.
  Interventions: Drug: IMG-007; Drug: Placebo

INTERVENTIONS:
Drug: IMG-007 — Participants will receive IMG-007 subcutaneously.
Drug: Placebo — Participants will receive a placebo subcutaneously.
  Arms: Placebo Crossover

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of different dose regimens of IMG-007, compared to placebo.

DETAILED DESCRIPTION:
A Phase 2b, multicenter, randomized, double-blind, placebo-controlled, parallel group study to assess the efficacy and safety profile of various dose regimens of IMG-007 in adult participants with moderate-to-severe active atopic dermatitis (AD) up to 52 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* Moderate-to-severe AD
* Documented history of inadequate response or lack of tolerability to a stable regimen of one or more topical treatment before the Screening visit, or for whom topical treatments are otherwise inadvisable
* Female participants who are not pregnant or breastfeeding and meet at least one of the following conditions: not of childbearing potential or of childbearing potential and agrees to use a highly effective method of contraception
* Male participants must agree to use a highly effective method of contraception
* EASI score ≥16
* vIGA-AD score ≥3
* ≥10% body surface area (BSA) of AD involvement
* Mean peak pruritus numerical rating scale ≥ 4 during 7-days before randomization

Key Exclusion Criteria:

* Positive hepatitis B, hepatitis C, or human immunodeficiency virus infection
* Evidence of active or latent tuberculosis (TB)
* History of untreated or inadequately treated TB infection
* Active infection requiring treatment with systemic antibiotics, antivirals, antifungals, antiparasitics or antiprotozoals
* Active unstable pruritic skin conditions in addition to AD that would interfere with the assessment of AD based on the investigator's clinical judgement
* Other conditions or laboratory abnormality that could increase the risk associated with study participation or could interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into the study
* Having received any of the specified therapies within the specified timeframe(s) prior to the Baseline visit

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Mean percent change from baseline in EASI at Week 20 | Baseline, Week 20

SECONDARY OUTCOMES:
Mean percent change from baseline in EASI at Week 16 | Baseline, Week 16
Proportion of participants achieving a ≥ 75% reduction in EASI (EASI-75) at Week 16 and Week 20, respectively | Week 16, Week 20
Proportion of participants achieving a vIGA-AD score of 0 (clear) or 1 (almost clear) and a ≥ 2-point reduction from baseline at Week 16 and Week 20, respectively | Week 16, Week 20
Incidence and severity of TEAE including treatment-emergent SAEs | Baseline, End of Study

CONTACTS AND LOCATIONS:
Locations (21):
- United States (15):
  - Antelope Valley Clinical Trials, Lancaster, California
  - Renstar Medical Research, Ocala, Florida
  - Palm Harbor Dermatology PA d/b/a TrueBlue Clinical Research, Tampa, Florida
  - Arlington Dermatology, Rolling Meadows, Illinois
  - Forest Hills Dermatology Group, Kew Gardens, New York
  - Inmagene Site 1, New York, New York
  - Vitality Clinical Trials LLC, Woodbury, New York
  - Darst Dermatology, Charlotte, North Carolina
  - Red River Research Partners, LLC, Fargo, North Dakota
  - ClinOhio Research Services LLC., Columbus, Ohio
  - Apex Clinical Research Center, Mayfield Heights, Ohio
  - Oregon Dermatology and Research Center, Portland, Oregon
  - Palmetto Clinical Trial Services, LLC, Anderson, South Carolina
  - Stryde Research-Epiphany Dermatology, Southlake, Texas
  - Dermatology of Seattle & Bellevue, Burien, Washington
- Canada (6):
  - Dr. Chin-ho-Hong Medical Inc., Surrey, British Columbia
  - Sudbury Skin Clinique, Greater Sudbury, Ontario
  - DermEdge Research, Mississauga, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Skinsense Medical Research, Saskatoon, Saskatchewan